CLINICAL TRIAL: NCT02309333
Title: Assessing the Impact of a Simplified Patient Care Strategy to Decrease Early Deaths In Acute Promyelocytic Leukemia (APL) By Maintaining A Database
Brief Title: Impact of a Simplified Patient Care Strategy to Decrease Early Deaths in Acute Promyelocytic Leukemia (APL) by Maintaining a Database
Status: Terminated | Type: Observational
Why Stopped: Previous principal investigators left institution
Sponsor: Emory University (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Principal Investigator, Martha Arellano, Principal Investigator, Emory University
Other Study IDs: IRB00067432; WINSHIP2488-13 (Other: Winship Cancer Institute)
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Leukemia, Promyelocytic, Acute
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute promyelocytic leukemia (APL) is a very rare type of leukemia. Because it is so rare, many doctors do not have experience treating it. APL has been shown to be curable most of the time. Unfortunately, some patients die early after they become sick with APL, sometimes even before starting treatment. The early period is from the time of diagnosis through the first treatments for the disease. This is approximately 30 days. Early deaths are often due to complications caused by of the effects of leukemia and the treatments of it. These complications may not be noticed quickly by doctors who don't have much experience with managing APL.

The purpose of this study is to collect information about the diagnosis and management of APL patients by review of their medical records. This information will be stored in a central database at Emory University. This data will be analyzed to discover the impact of increased physician knowledge of recommended management of APL. The goal is to reduce the events of early death of APL patients.

DETAILED DESCRIPTION:
The investigators propose to collect data on patients with APL treated predominantly across the states of Georgia and South Carolina but will also extend it to cover patients from neighboring states. The treatment will be as per the treating physician and would be standard of care and no new drugs or changes to standard of care are being proposed in educating the treating physicians.

This is a multi-center study. At the lead sites, patients will sign the consent form and data will be collected at those respective sites. The sites outside of Emory are centers in the catchment area that treat leukemia. The lead investigators are available around the clock to co-manage the APL patients.

The objective of the study is to collect data to assess for improvement in mortality at the primary centers as well as at the local treatment centers. This change in mortality would depend on educating the community physicians and nursing staff and requires regular visits both by the physicians and the nurse coordinator. The community hematologists/oncologists in the catchment area will be educated by sending emails from investigators at 3 month intervals to inform them of the high early death rate associated with APL. In addition, a brief pamphlet will be mailed to them once every 3 months as a reminder. The lead investigators in each state will make presentations in regional meetings, visit practices, and also call local practices. In addition, a nurse coordinator will be instrumental in calling upon nursing staff in outlying hospitals in the catchment area to apprise them of early deaths in APL and also make them aware of the study and resources available. This will be done aggressively during the first 6 months prior to initiating the trial and will be continued during the three-year study period.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of APL
* Positive t (15:17) by fluorescence in situ hybridization (FISH)
* Promyelocytic leukemia (PML)/retinoic acid receptor (RAR) alpha by polymerase chain reaction (PCR)

Exclusion Criteria:

* Only patients who refuse to provide consent will be excluded from the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with APL treated predominantly across the states of Georgia and South Carolina, as well as from neighboring states.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2014-11; Primary Completion 2016-11 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Mortality in the first month after diagnosis | 1 month after diagnosis

SECONDARY OUTCOMES:
Overall survival 18 months after accrual is completed | 18 months after accrual completion
Severity and duration of coagulopathy | 5 years from start of trial
  Assessment of the severity and duration of coagulopathy, including presence or absence of clinically evident bleeding or bruising, and laboratory data including prothrombin time, activated partial thromboplastin time, international normalized ratio (INR), D-dimer, and fibrinogen
Mortality with the severity and duration of coagulopathy | 5 years from start of trial
  Correlation of mortality with the severity and duration of coagulopathy
Bleeding and infections and length of stay in hospital | 5 years from start of trial
  Correlation of bleeding and infections and length of stay in hospital
Differentiation syndrome and length of hospital stay | 5 years from start of trial
  Correlation of differentiation syndrome (dyspnea, unexplained fever, weight gain, peripheral edema, unexplained hypotension, acute renal failure [ARF], congestive heart failure [CHF], pleuropericardial effusions and interstitial pulmonary infiltrates) and length of hospital stay
Safety by grade 3 or 4 toxicity | 5 years from start of trial
  Assessment of safety by grade 3 or 4 toxicity
Time to initiation of treatment from diagnosis | 5 years from start of trial
  Correlation of outcomes with time to initiation of treatment from diagnosis
Outcomes across different treatment centers | 5 years from start of trial
  Comparison of outcomes across different treatment centers.

CONTACTS AND LOCATIONS:
Overall Officials: Martha Arellano, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Medical University of South Carolina, Charleston, South Carolina
  - Gibbs Cancer Center and Research Institute, Spartanburg, South Carolina

REFERENCES:
- [Derived] Jillella AP, Arellano ML, Gaddh M, Langston AA, Heffner LT, Winton EF, McLemore ML, Zhang C, Caprara CR, Simon KS, Bolds SL, DeBragga S, Karkhanis P, Krishnamurthy SH, Tongol J, El Geneidy MM, Pati A, Gerber JM, Grunwald MR, Cortes J, Bashey A, Stuart RK, Kota VK. Comanagement Strategy Between Academic Institutions and Community Practices to Reduce Induction Mortality in Acute Promyelocytic Leukemia. JCO Oncol Pract. 2021 Apr;17(4):e497-e505. doi: 10.1200/OP.20.00395. Epub 2020 Oct 30. PMID 33125295